CLINICAL TRIAL: NCT01565304
Title: Evaluation of the Effectiveness of the POWER Through Choices Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MPR-06549-03
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy; Sexually Transmitted Infections
Keywords: Teen pregnancy; Sexually transmitted infections; Sexual risk behaviors
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POWER Through Choices (Experimental): 10-session group-based sexual education curriculum
  Interventions: Behavioral: POWER Through Choices
- Usual services (No Intervention): No intervention

INTERVENTIONS:
Behavioral: POWER Through Choices — 10-session group-based sexual education curriculum
  Arms: POWER Through Choices

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the POWER Through Choices (PTC) curriculum in increasing contraceptive use and delaying sexual initiation among youth living in group foster care homes.

DETAILED DESCRIPTION:
Youth in foster care are at especially high risk for teen pregnancy and associated sexual risk behaviors. The POWER Through Choices (PTC) program is a 10-session sexuality curriculum that aims to increase contraceptive use and delay sexual initiation by empowering youth to make healthy, positive choices about their sexual behaviors. This study uses a cluster randomized design to compare the effectiveness of PTC to usual programs and services provided to youth living in group foster care homes. Study participants will be youth living in group foster homes recruited in four locations: Kern County, CA; Cook County, IL; Baltimore County, MD; and Oklahoma (statewide). The study is being conducted as part of the national Evaluation of Adolescent Pregnancy Prevention Approaches funded by the Office of Adolescent Health in the U.S. Department of Health and Human Services.

ELIGIBILITY:
Inclusion Criteria:

* Resident of group foster care home

Exclusion Criteria:

* Pregnant or parenting

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1039 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Consistent contraceptive use | 12 months
Sexual initiation | 12 months

SECONDARY OUTCOMES:
Knowledge of contraceptive use and reproductive health | 6 months
Intentions to delay sexual initiation and unprotected sex | 6 months
Attitudes toward sexual activity and contraceptive use | 6 months
Scores on scale of self-efficacy to avoid sexual risk behaviors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roy Oman, PhD, Principal Investigator — University of Oklahoma; Sara Vesely, PhD, Principal Investigator — University of Oklahoma; Brian Goesling, PhD, Principal Investigator — Mathematica Policy Research
Locations (3):
- United States (3):
  - Kern County Superintendent of Schools, Bakersfield, California
  - Planned Parenthood of Maryland, Baltimore, Maryland
  - Oklahoma Institute for Child Advocacy, Oklahoma City, Oklahoma